CLINICAL TRIAL: NCT05223738
Title: Tissue Resident Memory T Cells in Early & Late Cases of Generalized Non-segmental Vitiligo
Brief Title: Resident Memory T Cells in Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Assistant Professor, Kasr El Aini Hospital
Other Study IDs: TRMvit
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to detect the presence and diversity of Tissue resident memory T cell populations in early and late cases of generalized non-segmental Vitiligo.

DETAILED DESCRIPTION:
* Written informed consent obtained from every participant.
* Detailed history taking including onset, course, duration of the disease, aggravating factors and received medications
* VASI score assessed in every patient.
* Patients photographed, divided into two groups early & late cases and 3 mm punch biopsies will be taken from perilesional and non lesional skin.
* Biopsies processed and stained for CD8 & CD69 in cases of early group, & late group and controls by immunofluorescence.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with Generalized non-segmental Vitiligo ( lesions in more than one anatomical site ).
* Both genders.
* Early group: onset less than or equal 6 months.
* Late group: onset more than 6 months

Exclusion Criteria:

* Localized or Segmental Vitiligo.
* Age < 14 years.
* Pregnant females
* Patient who received treatment of any type within the last 3 months for the late group.
* Patients with other skin diseases or immunosuppression

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Generalized Non-segmental Vitiligo
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
CD8+ immunofluorescence | 6months-1 year
  Number of Tissue resident Memory cells by positively stained by CD8+ in early and late generalized non segmental vitiligo patients
CD69+ immunofluorescence | 6months-1 year
  Number of Tissue resident Memory cells by positively stained by CD8+ in early and late generalized non segmental vitiligo patients
Double CD8+ and CD69+ immunofluorescence | 6months-1 year
  Number of Tissue resident Memory cells by double stained by CD8+ &CD 69+ in early and late generalized non segmental vitiligo patients
VASI | 6months-1 year
  Vitiligo Area and Severity index minimum 0 maximum 100, the larger the number the worse the condition

CONTACTS AND LOCATIONS:
Overall Officials: Hilal, Principal Investigator — Kasr El Ainy University Hospital, Faculty of medicine, Cairo University
Locations (1):
- Kasr El Ainy University hospital, Cairo, Egypt